CLINICAL TRIAL: NCT04921280
Title: Effectiveness of Internet-based Cognitive Behavior Therapy for Severe Health Anxiety in Clinical Psychiatry.
Brief Title: Effectiveness of ICBT for Severe Health Anxiety in Clinical Psychiatry.
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Volen Ivanov, Principal investigator, Karolinska Institutet
Other Study IDs: 2011/2091-31/3
Record Dates: First submitted 2021-05-04; First posted 2021-06-10 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Health Anxiety; Hypochondriasis; Illness Anxiety Disorder; Somatic Symptom Disorder; Severe Health Anxiety; Hypochondriacal Disorder, Unspecified
MeSH Terms: conditions — Hypochondriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Patients who have received treatment for severe health anxiety at the Internet Psychiatry Clinic, Psychiatry Southwest, Karolinska University Hospital Huddinge between April 2018 to April 2021.
  Interventions: Behavioral: Internet based Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Internet based Cognitive Behavioural Therapy — The treatment program consists of 12 chapters or "modules" spread over 12 weeks and contains written information, different exercises and weekly homework assignment. Patients get access to the CBT program via an internet portal and they have weekly contact with a licenced psychologist via encrypted email. Focus of the therapist support is to review the content of the weekly module, reinforce progress and engagement in therapy and assist with treatment difficulties. If needed, therapist can contact patients via telephone. Patients receive weekly reminders via SMS to login to the portal and fill out self-report measures.

SUMMARY:
The aim of this study is to evaluate the clinical effectiveness of internet-based cognitive therapy for severe health anxiety within regular psychiatric care.

A longitudinal cohort study will be conducted investigating 400 patients who have received ICBT for severe health anxiety between 2018-2020 in an outpatient psychiatric clinic providing Internet-based treatment.

The primary outcome measure will be the Short Health Anxiety Inventory, SHAI, and a within-group design with repeated measures will be used for primary analysis.

It is hypothesized that ICBT will be associated with a significant reduction in health anxiety as measured with SHAI, both after treatment and at six-month follow-up.

DETAILED DESCRIPTION:
Severe health anxiety is a prevalent disorder, leading to considerable distress and is associated with high societal costs. Internet-based cognitive behaviour therapy is a method to improve access to evidence-based psychological treatments and it has shown to be efficacious in the treatment of severe health anxiety in several randomized controlled trials. However, there is limited knowledge of its effectiveness and application in clinical psychiatric care.

The aim of this study is to evaluate the clinical effectiveness of internet-based cognitive therapy for severe health anxiety within regular psychiatric care.

The investigators will conduct at a cohort-study with a pretest-posttest design investigating consecutively recruited patients from May 2018 to April 2021 in an outpatient psychiatric clinic specialised in delivering ICBT. The treatment content has been successfully tested in previous efficacy studies and will be delivered during 13 weeks. The primary outcome measure will be the gold standard SHAI and a within-group design with repeated measures will be used in the primary analysis. It is estimated that 400 patients will receive treatment during this period and thus be included in the study, if consenting.

It is hypothesized that ICBT will be associated with a significant reduction in health anxiety as measured with SHAI, both after treatment and at six-month follow-up. The effect size is expected to be somewhat smaller than in research trials but still moderate to large (d > 0.5).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 16 years of age
* Living in Sweden
* Primary diagnosis of hypochondriasis according to ICD-10
* Able to read and write
* Have access to a computer or other device with an Internet connection
* If on medication, have a stable dose of psychotropic medication for 4 weeks prior to treatment
* Not having other psychiatric difficulties (e.g., ongoing substance abuse or a psychotic syndrome) that makes ICBT an unsuitable intervention

Exclusion Criteria:

* Patients with severe depression (clinician rated Montgomery-Asberg Depression Rating Scale- Self-Rated; MADRS-S and/or moderate to high risk of suicide in which monitoring is required
* Patients with low motivation, severe apathy, or difficulty concentrating
* Patients with psychosis
* Patients with untreated drug or alcohol problems
* Patients with reading and/or writing difficulties, including language difficulties;

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients will receive treatment at the Internet Psychiatry Clinic (www.internetpsykiatri.se), Psychiatry Southwest, Karolinska University Hospital Huddinge. Patient can either apply for treatment through self-referral or through referral from primary or psychiatric care. Self-referred patients will register for treatment through a public e-service portal for health care (i.e.Vårdguiden; 1177.se).
  Prior to treatment, patients will complete an online screening battery of self-report questionnaires and undergo an assessment by psychiatrists, or resident physicians supervised by psychiatrists.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
The short health anxiety inventory, SHAI | Change from baseline (week 0) to post-treatment (week 12)
  A 14-item self-report measure of health anxiety severity. Total scores on the scale range from 0 to 42 with higher scores indicating a worse outcome (more severe symptoms of health anxiety).

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale Self Rate, MADRS-S | Change from baseline (week 0) to post-treatment (week 12)
  A 10-item self-report measure of depressive symptoms. Total scores on the scale range from 0 to 54 with higher scores indicating a worse outcome (more severe depressive symptoms).
Generalised Anxiety Disorder 7-item scale, GAD-7 | Change from baseline (week 0) to post-treatment (week 12)
  A 7-item self-report measure of general anxiety symptoms. Total scores on the scale range from 0 to 21 with higher scores indicating a worse outcome (more symptoms of general anxiety).
EQ5D | Change from baseline (week 0) to post-treatment (week 12)
  A self-report measure of health-related quality of life.Total scores on the scale range from 0-1 with higher scores indicating a better outcome (more health and life quality). The questionnaire also includes a Visual Analog Scale (VAS) with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

CONTACTS AND LOCATIONS:
Overall Officials: Volen Ivanov, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- M46: Karolinska Universitetssjukhuset, Psykiatri Sydväst Stockholm, Huddinge, Sweden, 141 86, Stockholm, Sweden